CLINICAL TRIAL: NCT06098118
Title: Adapting a Mammography Decision Aid to Support Women Living in a Community Contaminated by Per- and Polyfluoroalkyl Substances (PFAS)
Brief Title: Adapting a Mammography Decision Aid to Support Women Living in a Community Contaminated by PFAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Christine M. Gunn, Assistant Professor, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00032987
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Screening
Keywords: per- and polyfluoroalkyl substances; breast cancer screening; decision aid; risk assessment
MeSH Terms: conditions — Progressive Encephalomyelitis with Rigidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid (Experimental): Participants will receive the adapted MyMammogram decision aid that includes environmental risk information.
  Interventions: Behavioral: MyMammogram decision aid

INTERVENTIONS:
Behavioral: MyMammogram decision aid — An online breast cancer screening decision aid that includes personalized risk assessment, information on benefits and risks of mammography screening, values clarification, outcome expectancies, and a summative document with participant responses.

SUMMARY:
This community-engaged research project will test an adapted online breast cancer screening decision aid to address the needs of women living in an area where environmental contamination has increased concern about breast cancer risk. It will provide novel data on individual experiences with breast cancer risk assessment and decisional determinants of screening choices in a community disproportionately impacted by industrial pollution.

DETAILED DESCRIPTION:
Environmental contamination is increasingly recognized as a critical driver of cancer disparities, and communities impacted by industrial pollution experience greater risk of cancer and higher cancer worry which complicates health decision making. Recently the National Academies of Science Engineering and Medicine (NASEM) released guidance suggesting that per- and polyfluoroalkyl substances (PFAS) are suggestively associated with breast cancer risk and that individuals with moderate to high blood concentrations of these chemicals should screen for breast cancer according to age and other risk factors as recommended by the US Preventive Services Task Force (USPSTF). Mammography screening guidelines for women in their 40s increasingly call for the use of risk assessment tools to guide screening initiation and imaging intervals (e.g. every year vs. every two years), but current tools do not address environmental risk factors that can contribute to breast cancer risk. This poses a particular challenge in communities where there is a real or perceived increased risk of breast cancer stemming from an environmental contamination concern. There are currently no decision tools tailored to help women living in such communities with their decisions about breast cancer screening. Therefore, the goal of the proposed work is to test an adapted online decision aid to incorporate environmental risk messaging to increase informed breast cancer screening decisions for women 40-49 years of age living in the greater Merrimack, New Hampshire area, where known and ongoing PFAS contamination exists. In partnership with Merrimack Citizens for Clean Water, we will distribute a community survey among screening-eligible women to test the new risk messaging within the decision aid (n=100) and establish acceptability in an open-label, single arm trial. The proposed research will contribute novel data on community-driven priorities for information about environmental contaminants that may affect breast cancer risk assessment and screening decisions.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 39-49
* No personal history of breast cancer,
* No mammogram in the prior 12 months
* Resident of Merrimack, Hillsborough, Rockingham or Bennington counties

Exclusion Criteria:

* History of breast cancer, ductal carcinoma in situ, lobular carcinoma in situ
* Cognitive impairment impeding the ability to provide informed consent

Ages: 39 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Acceptability | Within 1 day, post-intervention
  Acceptability e-scale,72 a 6-item measure for electronically-delivered interventions

SECONDARY OUTCOMES:
Knowledge | Immediately pre-intervention, within 1 day post-intervention
  10 Knowledge items summed to measure understanding of clinical screening, alternatives, main benefits/risks
Decisional Conflict | Immediately pre-intervention, within 1 day post-intervention
  The "SURE" measure, a 4-item validated checklist to assess decisional conflict, including benefits and risks of test
Screening self-efficacy | Immediately pre-intervention, within 1 day post-intervention
  10-item validated scale measuring self efficacy in obtaining mammography with summed score, range 5-50
Screening Intentions | Immediately pre-intervention, within 1 day post-intervention
  15-point validated scale measuring intentions and 1 decision question (yes/no/unsure)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Gunn, PhD, Principal Investigator — Dartmouth College, Geisel School of Medicine
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data that has been de-identified will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available after primary paper is published and for up to 3 years.

REFERENCES:
- [Derived] St Angelo M, Romano ME, Gallagher L, Gunn CM. Supporting informed decisions about breast cancer screening in communities with known environmental contamination: a pre-post study. Cancer Causes Control. 2025 Dec 27;37(1):11. doi: 10.1007/s10552-025-02100-5. PMID 41455034